CLINICAL TRIAL: NCT01880307
Title: Infliximab Top-down Study in Kids With Crohn's Disease
Brief Title: Infliximab Top-down in Pediatric Crohn
Acronym: ITSKids
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough study subjects
Sponsor: Erasmus Medical Center (Other)
Collaborators: University of Roma La Sapienza (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Lissy de Ridder, MD PhD, Pediatric gastroenterologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL39202.078.12; 2012-000645-13 (EudraCT Number); 2014-005702-37 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-18 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; pediatric; infliximab; top-down; ITSKids
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Top-down (Experimental): Infliximab and azathioprine; patients will receive 5 infliximab infusions of 5 mg/kg (IFX induction at week 0, 2 and 6, followed by 2 maintenance infusions every 8 weeks). IFX will be discontinued after 5 IFX infusions. Patients will also receive oral azathioprine 2-3 mg/kg, once daily as maintenance treatment.
  Interventions: Drug: Azathioprine; Drug: Infliximab
- Step-up (Active Comparator): Prednisolon and azathioprine; Patients will receive induction treatment with oral prednisolone 1 mg/kg (maximum 40 mg) once daily for 4 weeks, then tapering of prednisolone in 6 weeks until stop, and receive oral azathioprine 2-3 mg/kg, once daily as maintenance treatment.
  Interventions: Drug: Azathioprine; Drug: Prednisolon

INTERVENTIONS:
Drug: Azathioprine
  Other Names: Imuran
Drug: Infliximab
  Other Names: Remicade
  Arms: Top-down
Drug: Prednisolon
  Arms: Step-up

SUMMARY:
The purpose of this study is to determine whether a top-down treatment approach, prescribing infliximab and azathioprine at diagnose, yields better outcome in comparison to the usual step-up treatment approach, starting with prednison and azathioprine, in moderate-to-severe pediatric Crohn's disease (CD) patients.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to determine whether a top-down treatment approach, prescribing infliximab and azathioprine at diagnose, yields better outcome in comparison to the usual step-up treatment approach, starting with prednison and azathioprine, in moderate-to-severe pediatric Crohn's disease (CD) patients.

Sample size: We will include 100 (2 x 50) patients. With these numbers a difference of 60% and 85% (= 25) can be shown at a power of 80% (2-sided α 0.05; nQuery Advisor).

Study design: an international open-label randomised controlled trial Study population: Children (age 3-17 yrs) with new-onset, untreated, CD with moderate-to-severe disease activity Intervention: Patients will be randomised to either top-down IFX treatment or conventional step-up treatment.

Treatment arm 1: Top-down IFX treatment will consist of a total of 5 IFX infusions of 5 mg/kg (IFX induction at week 0, 2 and 6, followed by 2 maintenance infusions every 8 weeks) combined with oral azathioprine (AZA) 2-3 mg/kg once daily. AZA therapy will continue after the last IFX infusion to maintain remission.

Treatment arm 2: Step-up treatment will consist of standard induction treatment by oral prednisolone 1 mg/kg (maximum 40 mg) once daily for 4 weeks, followed by tapering in 6 weeks until stop. Prednisolone will be combined with oral AZA 2-3 mg, once daily, as maintenance treatment.

Main study parameters/endpoints: Clinical remission at 52 weeks without need for additional IBD related therapy or surgery. Secondary endpoints include clinical response, remission and mucosal healing at week 10 and 52, growth and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Children (age 3-17 years, both male and female) with new-onset, untreated CD with moderate-to-severe disease activity assessed by a wPCDAI >40 will be eligible for inclusion after a diagnosis of CD was made based on the Porto criteria.

Exclusion Criteria:

Patients with the following characteristics will be excluded: immediate need for surgery, symptomatic stenosis or stricture in the bowel due to scarring, active perianal fistulas, severe co-morbidity, severe infection such as sepsis or opportunistic infections, positive stool culture, positive Clostridium difficile assay, positive tuberculin test or a chest radiograph consistent with tuberculosis or malignancy, those already started with CD specific therapy.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical remission without need for additional CD related therapy or surgery | 52 weeks
  Clinical remission is defined as a Pediatric Crohn's Disease Activity Index (wPCDAI) score of less than 10 points

SECONDARY OUTCOMES:
Clinical response and remission rate | 10 weeks
  Response is defined by a decrease in PCDAI score above 15 points compared to baseline. Remission is PCDAI<10
Mucosal healing | 10 and 52 weeks
  Assessed by endoscopy (SES-CD) and/or fecal calprotectin (<100microgram/gram)
Growth | 10 and 52 weeks
  Change in height and BMI Z-scores, bone age and pubertal development
Therapy failure rates over time | 52 weeks
  Therapy failure: primary non-response, loss of response according to wPCDAI and medication intolerance
Cumulative therapy use | 52 weeks
Adverse events rates | 52 weeks
  Adverse events includes therapy side effects, disease complications (fistulas, abscesses, strictures, surgery, extra-intestinal manifestations)
Long-term yearly remission rates without need for additional CD related therapy or surgery | 260 weeks
Long-term yearly clinical remission, response and mucosal healing (calprotectin) rates | 260 weeks
Yearly number of flares | 260 weeks
Cumulative therapy use | 260 weeks
Adverse event rates | 260 weeks

OTHER OUTCOMES:
Pharmacokinetic properties of infliximab | 52 weeks
Identification of predictive biomarkers of therapy response | 52 weeks
Correlation between clinical disease activity, fecal calprotectin and endoscopic disease severity | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lissy Ridder, de, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Sapienza University, Rome, Italy
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- See also: Summary on Medicines for Children Research Network — http://www.mcrn.nl/index.php?option=com_content&view=article&id=143&Itemid=576